CLINICAL TRIAL: NCT04501952
Title: A Phase 3 Randomized, Double-Blind Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Remdesivir (GS-5734™) Treatment of COVID-19 in an Outpatient Setting
Brief Title: Study to Evaluate the Efficacy and Safety of Remdesivir (GS-5734™) Treatment of Coronavirus Disease 2019 (COVID-19) in an Outpatient Setting
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to study enrollment feasibility and changing needs of non-hospitalized participants. This decision is not based on efficacy or safety concerns.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-540-9012; 2020-003510-12 (EudraCT Number)
Expanded Access: NCT04323761 (Approved for marketing)
Record Dates: First submitted 2020-08-05; First posted 2020-08-06 (Actual); Results first posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — remdesivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Remdesivir (RDV) (Experimental): Participants will receive a single dose of intravenous (IV) RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2 and 3.
  Interventions: Drug: RDV
- Placebo (Placebo Comparator): Participants will receive IV placebo to match (PTM) RDV on Days 1 to 3.
  Interventions: Drug: Placebo to Match RDV

INTERVENTIONS:
Drug: RDV — Administered as an intravenous infusion
  Other Names: GS-5734™; Veklury®
  Arms: Remdesivir (RDV)
Drug: Placebo to Match RDV — Administered as an intravenous infusion
  Arms: Placebo

SUMMARY:
The primary objectives of this study are to evaluate the efficacy of remdesivir (RDV) in reducing the rate of of coronavirus disease 2019 (COVID-19) related hospitalization or all-cause death in non-hospitalized participants with early stage COVID-19 and to evaluate the safety of RDV administered in an outpatient setting.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent, (individuals ≥ 18 years of age) or assent (individuals ≥ 12 and < 18 years of age) prior to performing study procedures. Individuals age ≥ 18 years may be enrolled with the consent of a legal representative where permitted according to local law and approved nationally and by the relevant institutional review board (IRB) or independent ethics committee (IEC). For individuals ≥ 12 and < 18 years of age, a parent or legal guardian must be willing and able to provide written informed consent prior to performing study procedures
* Either:

  * Age ≥ 18 years (at all sites) or aged ≥ 12 and < 18 years of age weighing ≥ 40 kg (where permitted according to local law and approved nationally and by the relevant IRB or IEC with at least 1 pre-existing risk factor for progression to hospitalization (chronic lung disease, hypertension, cardiovascular or cerebrovascular disease, diabetes, obesity (body mass index ≥ 30), immunocompromised, chronic mild or moderate kidney disease, chronic liver disease, current cancer, or sickle cell disease)
  * Or aged ≥ 60 years
* Severe acute respiratory syndrome (SARS)-coronavirus (CoV)-2 infection confirmed by molecular diagnosis (nucleic acid (polymerase chain reaction (PCR) or antigen testing) ≤ 4 days prior to screening
* Presence of ≥ 1 symptom(s) consistent with COVID-19 for ≤ 7 days prior to randomization
* Not currently requiring hospitalization (hospitalization defined as ≥ 24 hours of acute care)

Key Exclusion Criteria:

* Participation in any other clinical trial of an experimental treatment and prevention for COVID-19
* Prior hospitalization for COVID-19
* Treatment with other agents with actual or possible direct antiviral activity against SARS-CoV-2 or administration of any SARS-CoV-2 (or COVID-19) vaccine
* Requiring oxygen supplementation

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (104):
- United States (92):
  - Arizona Liver Health, Chandler, Arizona
  - Arizona Clinical Trials, Tucson, Arizona
  - St Joseph Hospital Eureka, Eureka, California
  - St. Joseph Heritage Healthcare, Fullerton, California
  - Elevated Health, Huntington Beach, California
  - Ruane Clinical Research Group, Los Angeles, California
  - LA Universal Center, INC., Los Angeles, California
  - Mills Clinical Research, Los Angeles, California
  - Kaiser Permanente Northern California, Oakland, California
  - FOMAT Medical Research, Oxnard, California
  - UC Davis Health, Sacramento, California
  - Kaiser Permanente Northern California, 6600 Bruceville Road, Sacramento, California
  - Kaiser Permanente Northern California, 2025 Morse Ave, Sacramento, California
  - Kaiser Permanente Northern California, 1200 El Camino Real, San Francisco, California
  - Kaiser Permanente Northern California, 2425 Geary Blvd, San Francisco, California
  - UCSF Medical Center, San Francisco, California
  - Kaiser Permanente Northern California, 250 Hospital Parkway, Suite 850, San Jose, California
  - Kaiser Permanente Northern California, 2500 Merced St, San Leandro, California
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - Premiere Medical Center of Burbank, Inc, Toluca Lake, California
  - Kaiser Permanente Northern California, 975 Sereno Drive, Vallejo, California
  - New Hope Research Development DBA HCD, Whittier, California
  - Centura Health Porter Place, Denver, Colorado
  - Nuvance Health, Danbury, Connecticut
  - RecioMed Clinical Research Network, Boynton Beach, Florida
  - Midland Florida Clinical Research Center, LLC, DeLand, Florida
  - Invesclinic, Fort Lauderdale, Florida
  - Lawnwood Regional Medical Center, Ft. Pierce, Florida
  - Evolution Clinical Trials, Hialeah Gardens, Florida
  - Encore Medical Research, Hollywood, Florida
  - Advanced Pulmonary Research Institute, Loxahatchee Groves, Florida
  - L&C Professional Medical Research Institute, Miami, Florida
  - Laguna Clinical Research Associates, Miami, Florida
  - CTMD Research, Inc, Palm Springs, Florida
  - IMIC Inc, Palmetto Bay, Florida
  - Luminous Clinical Research - South Florida Urgent Care, Pembroke Pines, Florida
  - St. Josephs Comprehensive Research Institute, Tampa, Florida
  - AIDS Research and Treatment Center of the Treasure Coast, Vero Beach, Florida
  - Triple O Research Institute PA, West Palm Beach, Florida
  - Agile Clinical Research Trials, Atlanta, Georgia
  - Mercer University School of Medicine, Macon, Georgia
  - Infectious Disease Associates of Kansas City, P.C.Infectious Disease Associates of Kansas City, P.C., Burr Ridge, Illinois
  - Metro Infectious Disease Consultants, Burr Ridge, Illinois
  - NorthStar Medical Center, Chicago, Illinois
  - NorthShore University Healthsystem, Evanston, Illinois
  - Tulane University, New Orleans, Louisiana
  - Holy Cross Hospital, Inc., Baltimore, Maryland
  - University of Maryland Baltimore, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - South Shore Hospital, South Weymouth, Massachusetts
  - VA Boston Healthcare System, West Roxbury, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Onyx Research Institute, Flint, Michigan
  - Memorial Hospital of Gulfport, Gulfport, Mississippi
  - Metro Infectious Disease Consultants, Kansas City, Missouri
  - Quality Clinical Research Inc., Omaha, Nebraska
  - AB Clinical Trials, Las Vegas, Nevada
  - AXCES Research Group, Santa Fe, New Mexico
  - New York Presbyterian Hospital, Flushing, New York
  - Northwell Health, New Hyde Park, New York
  - Atrium Health Carolinas Medical Center, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Rosedale Infectious Diseases, Huntersville, North Carolina
  - Christ Hospital, Cincinnati, Ohio
  - Cherokee Nation WW Hastings Hospital, Tahlequah, Oklahoma
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Temple University, Philadelphia, Pennsylvania
  - Avera Research Institute, Sioux Falls, South Dakota
  - University of Tennessee Health Science Center, Knoxville, Tennessee
  - Central Texas Clinical Research, Austin, Texas
  - UT Physicians, Bellaire, Texas
  - Baylor University Medical Center, 700 Scott and White Dr., College Station, Texas
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Care United Research, LLC, Forney, Texas
  - VIP Trials, Harlingen, Texas
  - University of Texas, Houston, Texas
  - The Crofoot Research Center, Inc, Houston, Texas
  - Baylor University Medical Center, 1901 North McArthur Blvd, Irving, Texas
  - Laguna Clinical Research Associates, Laredo, Texas
  - Diagnostic Clinic of Longview - Center for Clinical Research, Longview, Texas
  - STAAMP Research, San Antonio, Texas
  - Sugar Lakes Family Practice, Sugar Land, Texas
  - Baylor University Medical Center, 2201 MacArthur Dr., Suite 100, Waco, Texas
  - ClinPoint Trials, Waxahachie, Texas
  - Intermountain Healthcare, Murray, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Providence Regional Medical Center Everett, Everett, Washington
  - Sound Medical Research, Port Orchard, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Providence Medical Research Center, Spokane, Washington
  - Wisconsin Corporation for Biomedical Research, Milwaukee, Wisconsin
- Denmark (5):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus N
  - Rigshospitalet, Copenhagen
  - Hvidovre Hospital, Hvidovre
  - Odense University Hospital, Odense
- Spain (3):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Clinic, Barcelona
  - Hospital Universitario Infanta Leonor, Madrid
- United Kingdom (4):
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - University College Hospital, London
  - St Mary's Hospital, London
  - Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Derived] Rodriguez L, Lee HW, Li J, Martin R, Han D, Xu S, Moshiri J, Peinovich N, Camus G, Perry JK, Hyland RH, Porter DP, Abdelghany M, Gotte M, Hedskog C. SARS-CoV-2 resistance analyses from the Phase 3 PINETREE study of remdesivir treatment in nonhospitalized participants. Antimicrob Agents Chemother. 2025 Feb 13;69(2):e0123824. doi: 10.1128/aac.01238-24. Epub 2024 Dec 19. PMID 39699245
- [Derived] Brown SM, Katz MJ, Ginde AA, Juneja K, Ramchandani M, Schiffer JT, Vaca C, Gottlieb RL, Tian Y, Elboudwarej E, Hill JA, Gilson R, Rodriguez L, Hedskog C, Chen S, Montezuma-Rusca JM, Osinusi A, Paredes R. Consistent Effects of Early Remdesivir on Symptoms and Disease Progression Across At-Risk Outpatient Subgroups: Treatment Effect Heterogeneity in PINETREE Study. Infect Dis Ther. 2023 Apr;12(4):1189-1203. doi: 10.1007/s40121-023-00789-y. Epub 2023 Apr 19. PMID 37074613
- [Derived] Grundeis F, Ansems K, Dahms K, Thieme V, Metzendorf MI, Skoetz N, Benstoem C, Mikolajewska A, Griesel M, Fichtner F, Stegemann M. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2023 Jan 25;1(1):CD014962. doi: 10.1002/14651858.CD014962.pub2. PMID 36695483
- [Derived] Gottlieb RL, Vaca CE, Paredes R, Mera J, Webb BJ, Perez G, Oguchi G, Ryan P, Nielsen BU, Brown M, Hidalgo A, Sachdeva Y, Mittal S, Osiyemi O, Skarbinski J, Juneja K, Hyland RH, Osinusi A, Chen S, Camus G, Abdelghany M, Davies S, Behenna-Renton N, Duff F, Marty FM, Katz MJ, Ginde AA, Brown SM, Schiffer JT, Hill JA; GS-US-540-9012 (PINETREE) Investigators. Early Remdesivir to Prevent Progression to Severe Covid-19 in Outpatients. N Engl J Med. 2022 Jan 27;386(4):305-315. doi: 10.1056/NEJMoa2116846. Epub 2021 Dec 22. PMID 34937145

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe and the United States. The first participant was screened on 18 September 2020. The last study visit occurred on 06 May 2021.
Pre-assignment Details: 630 participants were screened.
Groups:
- Remdesivir (RDV): Participants received a single dose of intravenous (IV) RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2 and 3.
- Placebo: Participants received IV placebo to match (PTM) RDV on Days 1 to 3.
Period: Overall Study
Arm/Group | Remdesivir (RDV) | Placebo
Started | 292 | 292
Completed | 266 | 272
Not Completed | 26 | 20
Not completed — Adverse Event | 0 | 3
Not completed — Investigator's Discretion | 0 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrew Consent | 5 | 4
Not completed — Lost to Follow-up | 7 | 2
Not completed — Randomized and Never Treated | 13 | 9

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who were randomized into the study and received at least 1 dose of study treatment.
Groups:
- Remdesivir: Participants received a single dose of IV RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2 and 3.
- Placebo: Participants received IV PTM RDV on Days 1 to 3.
- Total: Total of all reporting groups
Arm/Group | Remdesivir | Placebo | Total
Number analyzed (Participants) | 279 | 283 | 562
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50 (15.3) | 51 (14.8) | 50 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 138 | 269
  Male | 148 | 145 | 293
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted means local regulators did not allow collection of race information.
  Participants
    Race: American Indian or Alaska Native | 15 | 21 | 36
    Race: Asian | 6 | 7 | 13
    Race: Black | 20 | 22 | 42
    Race: Native Hawaiian or Pacific Islander | 1 | 0 | 1
    Race: White | 228 | 224 | 452
    Race: Other | 3 | 2 | 5
    Race: Not Permitted | 6 | 7 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted means local regulators did not allow collection of ethnicity information.
  Participants
    Ethnicity: Hispanic or Latino | 123 | 112 | 235
    Ethnicity: Not Hispanic or Latino | 146 | 158 | 304
    Ethnicity: Not Permitted | 10 | 13 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 264 | 267 | 531
  Denmark | 5 | 5 | 10
  United Kingdom | 3 | 1 | 4
  Spain | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Coronavirus Disease 2019 (COVID-19) Related Hospitalization (Defined as at Least 24 Hours of Acute Care) or All-Cause Death by Day 28
Description: The composite outcome of COVID-19 related hospitalization (defined as at least 24 hours of acute care) or all-cause death by Day 28 was derived by combining the available all-cause death and COVID-19 related hospitalization reported by the site. The first COVID-19 related hospitalization was used for the percentage of COVID-19 related hospitalization or all-cause death. The percentage of the composite outcome was from the Kaplan-Meier estimate.
Time Frame: Randomization up to Day 28
Population: Full Analysis Set included all participants who were randomized into the study and received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir | Placebo
Number analyzed (Participants) | 279 | 283
percentage of participants | 0.7 | 5.4
Statistical Analysis 1: Comparison: Remdesivir vs Placebo; Test type: Superiority; p = 0.0076, Regression, Cox; P-value was estimated using the Cox regression with baseline stratification factors as covariates; Hazard Ratio (HR) = 0.134, 95% CI 2-sided [0.031 to 0.586] — Hazard ratio and two-sided 95% confidence interval (CI) were estimated using the Cox regression with baseline stratification factors as covariates

2. Primary Outcome: Percentage of Participants Who Experienced Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug and/or any AEs leading to premature discontinuation of study drug.
Time Frame: First dose date up to last dose date (maximum: 3 days) plus 30 days
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir | Placebo
Number analyzed (Participants) | 279 | 283
percentage of participants | 42.3 | 46.3

3. Secondary Outcome: Percentage of Participants With COVID-19 Related Medical Visits Attended in Person by the Participant and a Health Care Professional (MAVs) or All-Cause Death by Day 28
Description: The composite outcome of COVID-19 related MAVs or all-cause death by Day 28 was derived by combining the available all-cause death and COVID-19 related MAVs reported by the site. The percentage of the composite outcome was from the Kaplan-Meier estimate.
Time Frame: Randomization up to Day 28
Population: Modified Full Analysis Set included all participants who were randomized into the study, and received at least 1 dose of study treatment, and enrolled under protocol amendment 2 or later.
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir | Placebo
Number analyzed (Participants) | 246 | 252
percentage of participants | 1.7 | 8.5
Statistical Analysis 1: Comparison: Remdesivir vs Placebo; Test type: Superiority; p = 0.0024, Regression, Cox; P-value was estimated using the Cox regression with baseline stratification factors as covariates; Hazard Ratio (HR) = 0.191, 95% CI 2-sided [0.065 to 0.555] — Hazard ratio and two-sided 95% CI were estimated using the Cox regression with baseline stratification factors as covariates

4. Secondary Outcome: Percentage of Participants Who Died by Day 28
Time Frame: Randomization up to Day 28
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir | Placebo
Number analyzed (Participants) | 266 | 274
percentage of participants | 0 | 0

5. Secondary Outcome: Percentage of Participants With COVID-19 Related Hospitalization at Day 28
Description: COVID-19 related hospitalization is defined as at least 24 hours of acute care derived by COVID-19 related hospitalization reported by the site. The percentage of the outcome and the corresponding 95% confidence interval were from Kaplan-Meier estimate.
Time Frame: Randomization up to Day 28
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir | Placebo
Number analyzed (Participants) | 279 | 283
percentage of participants | 0.7 [0.2 to 2.9] | 5.4 [3.3 to 8.7]

6. Secondary Outcome: Percentage of Participants With COVID-19 Related Hospitalization or All-Cause Death by Day 14
Description: The composite outcome of COVID-19 related hospitalization (defined as at least 24 hours of acute care) or all-cause death by Day 14 was derived by combining the available all-cause death and COVID-19 related hospitalization reported by the site. The first COVID-19 related hospitalization was used for the percentage of COVID-19 related hospitalization or all-cause death. The percentage of the composite outcome was from the Kaplan-Meier estimate.
Time Frame: Randomization up to Day 14
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir | Placebo
Number analyzed (Participants) | 279 | 283
percentage of participants | 0.7 | 5.4
Statistical Analysis 1: Comparison: Remdesivir vs Placebo; Test type: Superiority; p = 0.0076, Regression, Cox; P-value were estimated using the Cox regression with baseline stratification factors as covariates; Hazard Ratio (HR) = 0.134, 95% CI 2-sided [0.031 to 0.586] — [estimate comment as in outcome 3, analysis 1]

7. Secondary Outcome: Percentage of Participants With COVID-19 Related MAVs or All-Cause Death by Day 14
Description: The composite outcome of COVID-19 related MAVs or all-cause death by Day 14 was derived by combining the available all-cause death and COVID-19 related MAVs reported by the site. The percentage of the composite outcome was from the Kaplan-Meier estimate.
Time Frame: Randomization up to Day 14
Population: Participants in the modified Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir | Placebo
Number analyzed (Participants) | 246 | 252
percentage of participants | 0.8 | 8.0
Statistical Analysis 1: Comparison: Remdesivir vs Placebo; Test type: Superiority; p = 0.0019, Regression, Cox; P-value were estimated using the Cox regression with baseline stratification factors as covariates; Hazard Ratio (HR) = 0.100, 95% CI 2-sided [0.023 to 0.430] — [estimate comment as in outcome 3, analysis 1]

8. Secondary Outcome: Time-Weighted Average Change in Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV-2) Viral Load From Baseline to Day 7
Description: The time-weighted average change from baseline to study Day 7 (DAVG7) in SARS-CoV-2 viral load is defined as the time-weighted average between the first postbaseline value through the last available value up to Day 7 minus the baseline value in SARS-CoV-2 viral load (log10 copies/mL). DAVG7 is calculated using the trapezoidal rule and the area under the curve (AUC). For participants with data through days prior to Day 7, the time-weighted average change used data up to last available timepoint. If there was no postbaseline data, the participant was excluded from the analysis.
Time Frame: Baseline up to Day 7
Population: Participants in the Virology Analysis Set (all the participants who were randomized into the study, received at least 1 dose of study treatment, and had positive SARS-CoV-2 viral load at baseline) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/ mililiter (mL)
Arm/Group | Remdesivir | Placebo
Number analyzed (Participants) | 211 | 208
log10 copies/ mililiter (mL) | -1.24 (1.123) | -1.14 (1.099)
Statistical Analysis 1: Comparison: Remdesivir vs Placebo; Test type: Superiority; p = 0.4318, ANCOVA; P-value were from an ANCOVA model with baseline viral load as a covariate; Least Squares Mean = 0.07, 95% CI 2-sided [-0.10 to 0.24], Standard Error of Mean 0.09 — Least squares Mean (LSM), standard error (SE) and 95% CI were from an ANCOVA model with baseline viral load as a covariate

9. Secondary Outcome: Time to Alleviation (Mild or Absent) of Baseline COVID-19 Symptoms as Reported on the COVID-19-adapted Influenza Patient-Reported Outcome Plus Questionnaire (FLU-PRO Plus)
Description: The COVID-19-adapted FLU-PRO Plus is a questionnaire that assesses the severity of symptoms in participants with COVID-19 across six body systems: nose, throat, eyes, chest/respiratory, gastrointestinal, and body/systemic. Each domain scores range from 0 (symptom free) to 4 (very severe symptoms). A higher score indicates increased symptom severity. Alleviation is defined as symptom scores of 0 (absent) or 1 (mild). Time to alleviation of baseline COVID-19 symptoms is defined (in days) as: First Date of the two consecutive dates achieving alleviation - First dose Date + 1. If a participant had not achieved symptom alleviation at last FLU-PRO Plus assessment or early discontinuation of study, the participant was censored at last FLU-PRO Plus assessment date.
Time Frame: First Dose Date up to Day 14
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Placebo: Participants received IV placebo to match RDV on Days 1 to 3.
Arm/Group | Remdesivir | Placebo
Number analyzed (Participants) | 66 | 60
days | NA [10.0 to NA] — Not enough event to estimate Median and Inter-Quartile Range | NA [13.0 to NA] — Not enough event to estimate Median and Inter-Quartile Range
Statistical Analysis 1: Comparison: Remdesivir vs Placebo; Test type: Superiority; p = 0.2987, Log Rank; p-value was based on stratified log-rank test with baseline stratification factor as strata; Hazard Ratio (HR) = 1.405, 95% CI 2-sided [0.733 to 2.693] — [estimate comment as in outcome 3, analysis 1]

10. Secondary Outcome: Percentage of Participants With Worsening After Alleviation of Baseline COVID-19 Symptoms as Reported on the COVID-19-adapted FLU-PRO Plus Questionnaire
Description: The worsening after alleviation of baseline COVID-19 symptoms is defined as for a participant who has achieved alleviation of baseline COVID-19 symptoms, if symptom scored as 2 or higher at baseline is scored as 2 or higher postbaseline after achieved alleviation, or symptoms scored as 1 at baseline are scored as 1 or higher postbaseline after achieved alleviation. The COVID-19-adapted FLU-PRO Plus was used. It is a questionnaire that assesses the severity of symptoms in participants with COVID-19 across six body systems: nose, throat, eyes, chest/respiratory, gastrointestinal, and body/systemic. Each domain scores range from 0 (symptom free) to 4 (very severe symptoms). A higher score indicates increased symptom severity. Alleviation is defined as symptom scores of 0 (absent) or 1 (mild).
Time Frame: First dose date up to Day 28
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir | Placebo
Number analyzed (Participants) | 23 | 15
percentage of participants | 30.4 | 13.3

11. Secondary Outcome: Percentage of Participants Who Required Oxygen Supplementation by Day 28
Time Frame: Randomization up to Day 28
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir | Placebo
Number analyzed (Participants) | 279 | 283
percentage of participants | 0.4 | 1.8
Statistical Analysis 1: Comparison: Remdesivir vs Placebo; Test type: Superiority; p = 0.2163, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to 3 days plus 30 days; All-Cause Mortality: Randomization to the end of study (maximum: 59 days)
Description: Adverse Events: Safety Analysis Set included all participants who were randomized into the study and received at least 1 dose of study treatment; All-Cause Mortality: All Randomized Analysis Set included all participants who were randomized in the study.
Arm/Group | Remdesivir | Placebo
All-Cause Mortality (participants affected / at risk) | 0/292 | 1/292
Serious Adverse Events (participants affected / at risk) | 5/279 | 19/283
Other Adverse Events (participants affected / at risk) | 48/279 | 49/283
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Remdesivir (N=279) | Placebo (N=283)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Mitral valve prolapse (Cardiac disorders) | 0 | 1
Covid-19 (Infections and infestations) | 1 | 2
Covid-19 pneumonia (Infections and infestations) | 0 | 7
Pneumonia (Infections and infestations) | 2 | 3
Viral myocarditis (Infections and infestations) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Blood pressure inadequately controlled (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Remdesivir (N=279) | Placebo (N=283)
Nausea (Gastrointestinal disorders) | 30 | 21
Headache (Nervous system disorders) | 16 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/52/NCT04501952/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT04501952/SAP_001.pdf